CLINICAL TRIAL: NCT05981118
Title: Comparison of Post-Inflammatory Pigment Alteration After Psoriasis Treatment (PIPA - Dermavant)
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Dermavant Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00099131
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: ICD10 Code L40.9 for Psoriasis
MeSH Terms: interventions — tapinarof

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betamethasone dipropionate 0.05% (Active Comparator): The betamethasone dipropionate 0.05% cream group will be treated with betamethasone dipropionate 0.05% cream once daily on both legs until clear or up to 12 weeks.
  Interventions: Drug: Betamethasone dipropionate 0.05%
- Tapinarof (Active Comparator): The tapinarof group will be treated with 1% tapinarof cream applied once daily to both legs until clear or up to 12 weeks.
  Interventions: Drug: Tapinarof

INTERVENTIONS:
Drug: Betamethasone dipropionate 0.05% — 0.05% cream group will be treated once daily on both legs until clear or up to 12 weeks
  Arms: Betamethasone dipropionate 0.05%
Drug: Tapinarof — 1% tapinarof cream applied once daily to both legs until clear or up to 12 weeks
  Arms: Tapinarof

SUMMARY:
The purpose of this prospective study is to evaluate the degree of post-inflammatory pigmentation alteration on legs of study subjects treated with two different psoriasis treatments. Betamethasone dipropionate 0.05% cream is a high potency steroid that is commonly used to alleviate the inflammation of psoriasis. Tapinarof is another medication approved for psoriasis; tapinarof activates aryl hydrocarbon receptors to downregulate inflammatory cytokines (such as interleukin [IL]-17) which play a large role in psoriasis. Study subjects will be randomized to receive one of these medications and will be followed to monitor for PIPA. Photographs will be taken to help evaluate visual changes. The Taylor Hyperpigmentation scale will be used to grade the area and severity of hyperpigmentation and hypopigmentation; severity of erythema, burning, peeling, and dryness will also be recorded. This will allow us to understand the effects of two standard-of-care psoriasis medications to better treat patients.

DETAILED DESCRIPTION:
Subjects will be randomized to either of the two treatment groups (betamethasone dipropionate or tapinarof) and will be treated with that medication for until clear or up to 12 weeks . Photographs will be taken before and after treatment. The betamethasone dipropionate 0.05% cream group will be treated with betamethasone dipropionate 0.05% cream once daily on both legs until clear or up to 12 weeks. The tapinarof group will be treated with 1% tapinarof cream applied once daily to both legs until clear or up to 12 weeks.

Subjects will return every 4 weeks for evaluation. If disease recurs after clearing, treatment will be re-instituted.

Both groups will also be followed up at 1 and 4 weeks after end of treatment to monitor for PIPA and any other after-treatment effects.

Healthcare providers and patients may benefit from the information obtained during this study; study subjects may directly benefit from participation as they will be treated with standard treatments for psoriasis. We hope the information gathered will help healthcare providers better serve patients and identify psoriasis treatment after-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18+) with Fitzpatrick skin type 3 or higher who have been diagnosed with ICD10 code L40.9 for psoriasis between [dates] at Atrium Health Wake Forest Baptist Medical Center.
2. Stable on other therapies such as biologics for at least 3 months before randomization.

Exclusion Criteria:

1. Lack of a diagnosis of psoriasis (ICD10 code L40.9) or Fitzpatrick skin type below 3.
2. Pigmentary changes that in the opinion of the investigator would compromise the ability to assess the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Examine the degree of Post-inflammatory pigment alteration (PIPA) in both intervention Arms | Baseline to week 1
  Details regarding the area of pigmentation changes, intensity of hyper- or hypopigmentation, erythema, burning, and dryness will be assessed. PIPA will be assessed using the Taylor Pigmentation Scale
Examine the degree of Post-inflammatory pigment alteration (PIPA) in both intervention Arms | Week 1 to week 4
  Details regarding the area of pigmentation changes, intensity of hyper- or hypopigmentation, erythema, burning, and dryness will be assessed. PIPA will be assessed using the Taylor Pigmentation Scale
Examine the degree of Post-inflammatory pigment alteration (PIPA) in both intervention Arms | Week 4 to week 12
  Details regarding the area of pigmentation changes, intensity of hyper- or hypopigmentation, erythema, burning, and dryness will be assessed. PIPA will be assessed using the Taylor Pigmentation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States